CLINICAL TRIAL: NCT02988154
Title: Investigating the Efficacy of Simulation Curricula in Neurosurgical Education
Brief Title: Simulation Efficacy in Neurosurgical Education
Acronym: SENSE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Collaborators: University of Oxford (Other)
Responsible Party: Principal Investigator, A. Nimer Amr, Investigator, Johannes Gutenberg University Mainz
Other Study IDs: SimLab_SSP_01
Record Dates: First submitted 2016-12-06; First posted 2016-12-09 (Estimated); Last update posted 2017-01-20 (Estimated); Status verified 2017-01

CONDITIONS: Educational; Simulation; Hydrocephalus; Intraventricular Hemorrhage
Keywords: Medical education; simulation; neurosurgical education; Simulation laboratory; Ventricular drain
MeSH Terms: conditions — Hydrocephalus

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm A: Simulation training cohort: Recruits to Arm A undergo simulation training (computer simulation of the procedure, followed by simulation on a dead animal model), after which they will attempt to perform an EVD procedure on their own, on a 3D-printed skull model that we designed.
  Interventions: Other: Simulation training
- Arm B: ''See one, do one'' cohort: Recruits to Arm B will witness an EVD placement as performed by an experienced surgeon, after which they will attempt to perform an EVD procedure on their own, using the aforementioned 3D-printed skull model. This mimics the ''see one, do one'' paradigm prevalent in surgical training.
  Interventions: Other: ''See one, do one'' approach

INTERVENTIONS:
Other: Simulation training — Simulation training (computer simulation of the procedure, followed by simulation on a dead animal model).
  Groups: Arm A: Simulation training cohort
Other: ''See one, do one'' approach — The participants watch an experienced surgeon perform the EVD placement, after which the participants attempt to perform the procedure independantly on the skull model.
  Groups: Arm B: ''See one, do one'' cohort

SUMMARY:
This study aims to investigate the efficacy of simulation in neurosurgical training.

DETAILED DESCRIPTION:
This study aims to investigate the efficacy of simulation in neurosurgical training. This will be assessed using accuracy and speed tests in the placement of external ventricle drain catheters (EVDs). EVD placement is a relatively simple neurosurgical procedure aimed at inexperienced young trainees.

This study has two arms. The recruits are inexperienced trainees and/or interns and students who have never performed EVD placements before. The recruits are randomly assigned (using computer-based randomisation) to either Arm A or Arm B.

Recruits to Arm A undergo simulation training (computer simulation of the procedure, followed by simulation on a dead animal model), after which the recruits will attempt to perform an EVD procedure on their own, on a 3D-printed skull model that we designed.

Recruits to Arm B will witness an EVD placement as performed by an experienced surgeon, after the recruits will attempt to perform an EVD procedure on their own, using the aforementioned 3D-printed skull model. This mimics the ''see one, do one'' paradigm prevalent in surgical training.

The efficacy of the simulation training will be assessed using the following criteria:

i. Accuracy test:

The accuracy of the catheter placement is assessed in both arms and compared to investigate whether there is a difference in the accuracy of the catheter placement in both arms.

ii. Speed test:

The speed of catheter placement is assessed in both arms and compared to investigate whether there is a difference in the speed of the catheter placement in both arms.

iii. Subjective surveys

The researchers will gauge the extent of the trainees' confidence in their surgical skills and their satisfaction with their training before and after completion of the simulation training using a questionnaire to be designed for this purpose. The trainees will assess their own familiarity with and confidence in the procedure using a scale from 0 ("not familiar with the procedure", "I have no confidence in being able to perform this procedure independently") to 10 ("I am an expert at this procedure", "I am able to perform this procedure independently with complete confidence"). This data will be collected and input into a statistical software (Statistical Lab v. 3, CeDiS) to analyse the difference (if any) in the trainees' familiarity with the procedures and their confidence in being able to perform them in both arms.

ELIGIBILITY:
Inclusion Criteria:

* never performed EVD placements before

Exclusion Criteria:

* any surgical experience with EVD placement

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: The recruits to the study are inexperienced surgical trainees and/or interns and students who have never performed EVD placements before.
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-01 (Estimated)

PRIMARY OUTCOMES:
Accuracy of catheter placement | immediately upon completion of the procedure
  The placement of the catheter will be analysed by blinded assessors. Outcome: is the catheter in the ventricle (yes/no).
Speed of performing the procedure | immediately upon completion of the procedure
  The time needed to complete the procedure will be recorded in seconds by blinded assessors.

SECONDARY OUTCOMES:
Subjective survey | To be taken immediately before and immediately after performing the EVD insertion

CONTACTS AND LOCATIONS:
Overall Officials: Alexander L Green, MD, Study Director — University of Oxford
Locations (1):
- University of Mainz / Department of Neurosurgery, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No